CLINICAL TRIAL: NCT02632929
Title: Prevention of Amputation in a High Risk Population With Comprehensive Care and Amniotic Tissue
Brief Title: Prevention of Amputation in Diabetic Foot Ulcers Using Amniotic Tissue
Status: Completed | Type: Observational
Sponsor: Boise VA Medical Center (U.S. Federal Agency)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Margaret Doucette, Director, Physical Medicine and Rehabilitation, Boise VA Medical Center
Other Study IDs: 00816
Record Dates: First submitted 2015-12-14; First posted 2015-12-17 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcer
Keywords: foot ulcer, diabetic; wound healing; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic Foot Ulcers at Amputation Risk: Patients at high risk for limb amputation from a diabetic foot ulcer will be treated with comprehensive, interdisciplinary approach (usual care) in combination with early application of advanced therapy; dehydrated human amniotic membrane allografts (AMNIOEXCEL®, Derma Science, Princeton, New Jersey).

SUMMARY:
The purpose of this study is to see whether the use of AMNIOEXCEL® improves healing and reduces the need to cut off all or part of a leg (amputation) in high-risk patients who have diabetes and foot sores (also sometimes called ulcers or wounds).

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the effectiveness of comprehensive, interdisciplinary approach (usual care) in combination with early application of advanced therapy; dehydrated human amniotic membrane allografts (AMNIOEXCEL®, Derma Science, Princeton, New Jersey) in healing and preventing amputation in high risk patients with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes
* Ulcer anywhere on the foot
* Moderate to high risk for amputation according to Prevention of Amputation for Veterans Everywhere (PAVE) and the Society for Vascular Surgery Lower Extremity Threatened Limb (SVS WIfI) classification system (WIFi) criteria

Exclusion Criteria:

* Inability or unwillingness to travel to Boise VA for clinic visits
* Enrolled in Hospice
* Have known or expected malignancy of foot ulcer
* Are or planning to become pregnant
* Signs of progressive gangrene, limb-threatening infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diabetic foot ulcer referred to the High Risk Foot Clinic at Boise VAMC who meet the inclusion criteria, and are willing and able to participate will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05-30; Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Limb salvage | One month past wound healing
  All subjects will be seen weekly/biweekly by the study team until the point of definitive wound closure (epithelialization) and the subject has the ability to progress weight bearing and ambulation.

SECONDARY OUTCOMES:
effective wound healing | One month past wound healing
  Early application of amniotic tissue and multidisciplinary team comprehensive care on diabetic foot ulcers with a high risk for amputation

OTHER OUTCOMES:
Diabetic Foot Ulcer Quality of life Short Form survey | Comparison of patient's perception at enrollment, wound heal, one month, and 2-4 months after the wound is healed.
  Quality of life measured at enrollment in study, at wound healed, one month post-healed, and 2-4 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Doucette, D. O., Principal Investigator — Boise VAMC; Kattie B Payne, PhD, RN, MSN, Study Director — Boise VAMC
Locations (1):
- Boise VAMC, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study.

REFERENCES:
- [Background] Mills JL Sr, Conte MS, Armstrong DG, Pomposelli FB, Schanzer A, Sidawy AN, Andros G; Society for Vascular Surgery Lower Extremity Guidelines Committee. The Society for Vascular Surgery Lower Extremity Threatened Limb Classification System: risk stratification based on wound, ischemia, and foot infection (WIfI). J Vasc Surg. 2014 Jan;59(1):220-34.e1-2. doi: 10.1016/j.jvs.2013.08.003. Epub 2013 Oct 12. PMID 24126108
- [Background] Abetz, L., Sutton, M., Brady, L., McNulty, P., Gagnon, D. The Diabetic Foot Ulcer Scale (DFS): a quality of life instrument for use in clinical trials. Pract Diab Int July/August 2002 Vol 19 No. 6
- [Background] Bann CM, Fehnel SE, Gagnon DD. Development and validation of the Diabetic Foot Ulcer Scale-short form (DFS-SF). Pharmacoeconomics. 2003;21(17):1277-90. doi: 10.2165/00019053-200321170-00004. PMID 14986739
- [Derived] Doucette M, Payne KM, Lough W, Beck A, Wayment K, Huffman J, Bond L, Thomas-Vogel A, Langley S. Early Advanced Therapy for Diabetic Foot Ulcers in High Amputation Risk Veterans: A Cohort Study. Int J Low Extrem Wounds. 2022 Jun;21(2):111-119. doi: 10.1177/1534734620928151. Epub 2020 Jun 22. PMID 32567415